CLINICAL TRIAL: NCT03631498
Title: Apoptosis and Tissue Destruction in Gingival Tissues of Smoker and Non-smoker Periodontitis Patients
Brief Title: Apoptotic Changes in Gingiva Caused by Smoking
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hatice Balci Yuce, Principal investigator, Tokat Gaziosmanpasa University
Other Study IDs: Ozkan
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Smoking; Chronic Periodontitis
Keywords: smoking; hypoxia; apoptosis; chronic periodontitis
MeSH Terms: conditions — Smoking; Chronic Periodontitis; Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Gingival tissue biopsy samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy individuals: Gingival biopsies of healthy individuals who were never-smokers and had no systemic or oral disease or condition.
- periodontitis patients: Gingival biopsies of periodontitis patients who were never-smokers and had no systemic disease or condition.
- Healthy smokers: Gingival biopsies of healthy individuals who were smokers but no systemic or oral disease or condition.
- Smokers with periodontitis: Gingival biopsies of periodontitis patients who were smokers but no systemic disease or condition.

SUMMARY:
Smoking is a major environmental risk factor associated with common forms of human chronic periodontitis. The aim of the present study was to evaluate apoptotic tissue alterations and tissue destruction in smoker and non-smoker chronic periodontitis patients and healthy individuals. The investigators of the study suggest that smoking decrease tissue quality and increase inflammation level in gingival tissues in both healthy individuals and periodontitis patients. One possible mechanism for this is suggested to be increased apoptosis.

DETAILED DESCRIPTION:
Periodontal disease disrupts soft tissue metabolism in the gingiva through a decrease in the production of collagen, the quality, and quantity of the connective tissue. The etiology and pathogenesis of chronic periodontitis are mostly revealed, however, the mechanism of environmental factors such as smoking yet to be clarified. Major consequences of smoking in gingival tissues are suggested to be the reduction in neutrophil and fibroblast function, decreased immunoglobulin G production, increased periodontal pathogen bacteria prevalence, difficulty in eliminating pathogens with mechanical therapy, and reduction in growth factor production. In the present study, markers of tissue destruction, matrix metalloproteinase-8 and tissue inhibitor of matrix metalloproteinase-1, hypoxia markers, vascular endothelial growth factor and hypoxia-inducible factor and apoptotic markers, bax, bcl-2, and caspase-3 were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 30 to 45,
* the existence of at least 20 functioning teeth,
* systemical health,
* no antibiotic use within 6 months,
* no periodontal therapy within 6 months,
* no pregnancy or lactation,
* no drug use, in addition; for the smokers existence of the smoking condition for at least five years.

Exclusion Criteria:

* Patients younger than 30 older than 50 years old,
* the absence of occlusion,
* drug use,
* pregnancy/lactation,
* previous antibiotic use,
* previous periodontal therapy,
* the existence of any systemical disease.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals who were either smokers or non-smokers, chronic periodontitis patients who were either smokers or non-smokers older than 30 years old and younger than 50 years old were enrolled. The age was specifically chosen because aging changes periodontal and gingival tissues independently of other variables. Any possible factor which might alter connective tissue metabolism were excluded.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Fibroblast and total inflammatory cell counts | Biopsies were obtained a day after initial examinations, histological analysis were performed 2 weeks after.
  Fibroblast and total inflammatory cell counts in the groups were determined in a standardized 1000 micrometer square area with histomorphometric evaluation.

SECONDARY OUTCOMES:
Apoptotic markers | Biopsies were obtained a day after initial examinations, histological analysis were performed 2 weeks after
  Apoptotic and anti-apoptotic proteins and enzymes related to apoptosis were evaluated via immunohistochemistry.
Hypoxia and tissue destruction markers | Biopsies were obtained a day after initial examinations, histological analysis were performed 2 weeks after
  Vascular endothelial growth factor and hypoxia-inducible factor as hypoxia markers and matrix metalloproteinase and it inhibitor as destruction markers were evaluated via immunohistochemistry.

CONTACTS AND LOCATIONS:
Overall Officials: HATİCE BALCI YÜCE, PhD, Principal Investigator — Gaziosmanpasa University
Locations (1):
- Gaziosmanpasa University Faculty of Dentistry, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided